CLINICAL TRIAL: NCT01705626
Title: Screening for the Transthyretin-Related Familial Amyloidotic Polyneuropathy (TTR-FAP): An International, Multicenter, Epidemiological Protocol
Brief Title: Screening for the Transthyretin-Related Familial Amyloidotic Polyneuropathy (TTR FAP)
Acronym: TRAP2-1
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: TRAP 08-2012
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Polyneuropathy, Amyloid; Neuropathic Pain; Cardiac Failure; Orthostatic Hypotension; Gastrointestinal Disorders
Keywords: Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy; TTR FAP; Biomarker
MeSH Terms: conditions — Amyloid Neuropathies; Neuralgia; Heart Failure; Hypotension, Orthostatic; Gastrointestinal Diseases; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with small fiber polyneuropathy no obvious etiology: Participants aged between 18 and 85 years, diagnosed with small fiber polyneuropathy of no obvious etiology, without diagnosis of alcoholism and not undergoing chemotherapy for cancer

SUMMARY:
An International, multicenter, epidemiological observational study investigating the prevalence of Transthyretin-Related Familial Amyloidotic Polyneuropathy (TTR-FAP) in participants with small fiber polyneuropathy of no obvious etiology.

DETAILED DESCRIPTION:
Transthyretin-related Familial Amyloid Polyneuropathy (TTR-FAP) is an autosomal dominant, progressive neurodegenerative disease, with fatal outcome occurring within ten years after onset. Familial amyloid polyneuropathy (FAP) associated with mutations in the transthyretin (TTR) gene is the most common form of genetic amyloidosis. It accounts several thousand cases worldwide, with Val30Met mutation identified in most patients and with endemic foci in Portugal, Sweden and Japan.

TTR FAP is caused by the systemic deposition of amyloidogenic variants of the transthyretin protein ((Ttr) in the extra-cellular space of tissues and result in disruption of organ function.The typical presentation of TTR-FAP is a progressive sensory-motor polyneuropathy, which usually begins with loss of thermal and pain sensation in the feet, slowly ascends up the limbs and is associated with variable autonomic disturbances and extra-neurological manifestations (especially a cardiomyopathy).

The goal of the TRAP2.1 Study is to investigate the prevalence of Transthyretin-Related Familial Amyloidotic Polyneuropathy (TTR-FAP) in a cohort of 500 subjects with small fiber polyneuropathy of no obvious etiology, based on the subject's clinical presentation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* The participant is aged between 18 and 85 years of age
* The participant is diagnosed with small fiber polyneuropathy of no obvious etiology
* The participant has no diagnosis of alcoholism, according to International Guidelines
* The participant has not undergone chemotherapy for carcinoma

Exclusion Criteria:

* Inability to provide informed consent
* The participant is younger than 18 years or older than 85 years of age
* The etiology of the small fiber polyneuropathy is clearly determined
* The participant has a diagnosis of alcoholism, according to International Guidelines
* The participant has undergone chemotherapy for carcinoma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with small fiber polyneuropathy of no obvious etiology.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Epidemiological analysis of prevalence of the TTR FAP in participants with small fiber polyneuropathy of no obvious etiology. | 3 years
  Dry Blood Spot (DBS) samples will be genetically validated via combination of Next-Generation Sequencing (the mutation will be confirmed by Sanger sequencing) and the Multiplex ligation-dependent probe amplification (MLPA) of TTR gene

SECONDARY OUTCOMES:
Establishment of a biomarker in TTR-positive cohort | 3 years
  Samples carrying a mutation in the TTR gene will be biochemically analyzed via liquid chromatography multiple reaction monitoring MS and compared with a merged control cohort, in order to establish TTR mutation-specific biomarker/s.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmgH
Locations (11):
- Klinikum Wels-Grieskirchen GmbH, Abteilung für Neurologie, Wels, Austria
- Hungary (2):
  - University of Pécs, Department of Neurology, Pécs
  - University of Szeged, Department of Neurology, Szeged
- University Hospital Skopje, Department of Neurology, Skopje, North Macedonia
- Jagiellonian University Medical College, Department of Neurology, Krakow, Poland
- Serbia (4):
  - Clinical Hospital Center Zvezdara, Department of Neurology, Belgrade
  - University of Belgrade, Clinical Center of Serbia, Neurology Clinic, Neuropathy Center, Belgrade
  - Clinical Center Niš, Department of Neurology, Niš
  - General Hospital "Dr. Djordje Joanović", Zrenjanin
- Spain (2):
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Donostia, San Sebastián

IPD SHARING:
Plan to Share IPD: Undecided